CLINICAL TRIAL: NCT07169149
Title: Study of the Prevalence and Patterns of Drug Resistance of Mycobacterium Tuberculosis Using GeneXpert (MTB/RIF) and Xpert (MTB/XDR) Assays
Brief Title: Study About Drug Resistance of Mycobacterium Tuberculosis
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Omnia Abdelazim Mohamed, chest specialist, Sohag University
Other Study IDs: Soh-Med-25-8---3MD
Record Dates: First submitted 2025-08-19; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary and Extra- Pulmonary Tuberculosis (TB)
MeSH Terms: conditions — Tuberculosis, Extrapulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tuberculosis is a major cause of ill health and one of the leading causes of death worldwide. Early, rapid and accurate diagnosis of all TB patients and prompt treatment with any form of drug-susceptible or drug resistant TB is fundamental. Identifying the pattern of drug resistance will ensure that the most effective therapy can be selected. The aim of this study is to assess the prevalence and patterns of drug resistance of mycobacterium tuberculosis and to detect the possible risk factors associated with resistant cases.

ELIGIBILITY:
Inclusion Criteria:

* geneXpert positive patients in pulmonary and extrapulmonary cases

Exclusion Criteria:

* age below 12 years

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients with geneXpert positive samples whether rifampicin resistant or sensitive
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Detection of number of cases resistant to Rifampicin and other anti- TB drugs | within 6 months of starting treatment
  Using of GeneXpert (MTB/RIF) and Xpert (MTB/XDR) assays to detect resistance to Rifampicin and other anti -TB drugs among TB positive cases

SECONDARY OUTCOMES:
Detection of common Risk factors associated with resistant cases | within 6 months of starting treatment coarse
  collection of (in common) data among cases to detect risk factors associated with drug resistance e.g is drug resistance more common in diabetic patients?, is resistance more common among drug addict patients? , also is there common co-morbid conditions among resistant cases

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided